CLINICAL TRIAL: NCT02238886
Title: RADICAL CYSTECTOMY, NUTRITION AND CONVALESCENCE: CAN GOAL-DIRECTED POSTOPERATIVE NUTRITIONAL THERAPY REDUCE THE CONVALESCENCE PERIOD FOR PATIENTS UNDERGOING RADICAL CYSTECTOMY (RC)?
Brief Title: Radical Cystectomy, Nutrition and Convalescence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Line Noes Lydom, Clinical nurse specialist, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-2-2011-114
Record Dates: First submitted 2014-09-05; First posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Urinary Bladder Neoplasms; Cystectomy; Bladder Cancer
Keywords: Quality of Life; Enteral nutrition; Nutrition Therapy; Parenteral nutrition, total
MeSH Terms: conditions — Urinary Bladder Neoplasms; Hyperphagia

ARMS (2):
- Parenteral nutrition (Experimental): Patients receives a goal-directed nutritional intervention combining oral intake and parenteral nutrition
  Interventions: Dietary Supplement: Parenteral nutrition. SMOFKABIVEN infusion in central vene. Fresenius Kabi
- Standard treatment (No Intervention): patients receives a standard nutritional strategy of resting the bowel till clear signs of bowel recovery and feeding orally after bowel recovery

INTERVENTIONS:
Dietary Supplement: Parenteral nutrition. SMOFKABIVEN infusion in central vene. Fresenius Kabi
  Arms: Parenteral nutrition

SUMMARY:
The purpose of this study is to determine whether a goal directed nutritional intervention can reduce the convalescence period for patients undergoing radical cystectomy (RC).

The aim is to examine the effect on quality of life of a standard nutritional strategy of resting the bowel till clear signs of bowel recovery and feeding orally after bowel recovery versus a goal-directed nutritional intervention combining oral intake and parenteral nutrition, in patients undergoing RC.

DETAILED DESCRIPTION:
The study is a randomized controlled trial. Inclusion criteria: Bladder cancer, ability to give an informed consent. Exclusion criteria: Previous radiation therapy at the pelvic area, ureterocutaneostomy or robot-assisted surgery. The intervention aims to secure that 75% of the patient's total energy and protein needs are met during hospitalization.

Primary outcome: Quality of Life, using the EORTC QLQ-C30 and BLM30 questionnaire. Secondary outcomes: Body-weight, Hand Grip strength, biochemical measures, length of hospital stay, time to bowel recovery. The follow-up period is 12 weeks. Statistical analysis is performed in collaboration with a statistician.

ELIGIBILITY:
Inclusion Criteria:

* Bladder cancer
* Ability to give an informed consent

Exclusion Criteria:

* Previous radiation therapy at the pelvic area
* Ureterocutaneostomy
* Robot-assisted surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Health related quality of life (HRQoL) using the EORTC QLQ-C30 and BLM30 (one combined questionnaire) | meassured pre-operatively + 6 and 12 weeks following surgery
  Change from baseline HRQoL at 6 and 12 weeks following surgery

SECONDARY OUTCOMES:
Body weight | preoperatively, 6 and 12 weeks postop
  Change from baseline weight at 6 and 12 weeks following the date of surgery
hand grip strength | pre-operatively, 6 days and 6 weeks postop
  Change from baseline hand grip strength at 6 days and 6 weeks following the date of surgery
length of hospital stay | 12 week follow-up
Time to bowel recovery | 12 week follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Dep. of Urology. University Hospital Rigshospitalet, Copenhagen Denmark, Copenhagen, Denmark